CLINICAL TRIAL: NCT07170163
Title: Navigating the Transition to Adulthood: A Dual Language Mobile App for Latino Youth With ASD and Their Families
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Antonio Pagan, Post Doctoral Fellow, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-25-0519; 1R03HD119485 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: mHealth app
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ¡Iniciando! mHealth App (Experimental)
  Interventions: Behavioral: ¡Iniciando! mHealth App

INTERVENTIONS:
Behavioral: ¡Iniciando! mHealth App — Participants will undergo 12 weekly, 1-hour virtual group sessions (separate for young adults and parents) and weekly, 30-minute individual virtual coaching sessions for young adults (which parents may attend as appropriate). Participants will also engage with the ¡Iniciando! app modules before and after their virtual group meetings. Throughout the approximately three-month study period, participants will complete (e.g., usability, satisfaction, adherence, app usage data).

SUMMARY:
The purpose of this study is to determine useability and satisfaction characteristics,product usage data,methodological feasibility parameters and feasibility metrics of the mHealth app adapted intervention on the mental health, quality of life, and adaptive functioning of Latino transition aged young adults with ASD and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Latino young adults with ASD ASD with a score of 15 or greater on the Social Communication Questionnaire-Lifetime (SCQ-L)
* meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR), criteria for ASD based on a DSM-5-TR ASD symptom checklist
* previous diagnosis of ASD from a licensed mental health or medical professional(f they have not been diagnosed by a licensed mental health or medical professional, a complete a diagnostic evaluation will be conducted, using semi-structured interviews, questionnaires, the autism diagnostic interview-revised (ADI-R), and the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) to confirm ASD diagnosis)
* above the "moderate" cut off for symptoms of anxiety or depression( Depression and anxiety symptoms will be assessed via the Patient Health Questionnaire-9 (PHQ-9) and the Generalized Anxiety Disorder-7 (GAD-7)
* Spanish-speaking parents

Exclusion Criteria:

* low intelligence quotient (IQ) score (Verbal IQ < 70) on the verbal IQ on Kaufman Brief Intelligence Test Second Edition (KBIT-2)
* psychotic as determined by the Structured clinical interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM5): Research Version (SCID-5-RV), or are actively suicidal with an active plan.
* substance abuse

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited | end of study (about 3 months after baseline)
Source of participants | end of study (about 3 months after baseline)
  Participants maybe recruited from the following :
  UTHealth Houston Community Health Workers Social Media advertisements Private clinics
Time taken for recruitment of participants | end of study (about 3 months after baseline)
Number of participants that completed the study | end of study (about 3 months after baseline)
Usability as measured by the User Version of the Mobile Application Rating Scale (uMARS) | end of study (about 3 months after baseline)
  This is a 20 item questionnaire and each item is rated on a 5-point Likert scale, scores range from 1(inadequate) to 5(excellent) with higher scores indicating better usability.
Usability as Measured by the System Usability Scale (SUS) | end of study (about 3 months after baseline)
  The System Usability Scale (SUS) is a validated 10-item questionnaire . Each item is rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Scores are converted to a total SUS score ranging from 0 to 100, with higher scores indicating better usability. A score above 68 is generally considered above average usability.
Differences in outcome expectancy as assessed by the treatment credibility scales | end of study (about 3 months after baseline)
  this is a 6 item questionnaire and each is scored from 1-9, maximum score would be 54, higher score indicating better outcome
Treatment Adherence as assessed by the number of completed sessions | end of study (about 3 months after baseline)
Treatment Adherence as assessed by the homework completion rate | end of study (about 3 months after baseline)
Treatment Adherence as assessed by the number of participants that drop out | end of study (about 3 months after baseline)
Treatment Adherence as assessed by the time spent on homework | end of study (about 3 months after baseline)
Time-used on the mHealth app | end of study (about 3 months after baseline)
Percentage of modules completed on the mHealth app | end of study (about 3 months after baseline)
Frequencies of goal setting on the mHealth app | end of study (about 3 months after baseline)
Acceptability of Intervention as assessed by the Acceptability of Intervention Measure (AIM | end of study (about 3 months after baseline)
  This is a 4 item questionnaire and each is scored form 1( completely disagree) to 5 (completely agree) for a maximum score of 20, higher score indicating better outcome
Intervention Appropriateness as assessed by the Intervention Appropriateness Measure (IAM) | end of study (about 3 months after baseline)
  This is a 4 item questionnaire and each is scored form 1( completely disagree) to 5 (completely agree) for a maximum score of 20, higher score indicating better outcome
Feasibility of Intervention as assessed by the Feasibility of Intervention Measure (FIM) | end of study (about 3 months after baseline)
  This is a 4 item questionnaire and each is scored form 1( completely disagree) to 5 (completely agree) for a maximum score of 20, higher score indicating better outcome

SECONDARY OUTCOMES:
Change in depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) for depressive symptoms | baseline (+/-1 month), 6 weeks later (+/-1 month), and 12 weeks later ((+/-1 month)
  This is a 9 item questionnaire and each is scored from 0(not at all) to 3(nearly every day) for a maximum score of 27, higher number indicating worse outcome
Change in anxiety as assessed by the Generalized Anxiety Disorder-7 (GAD-7) for anxiety symptoms | baseline (+/-1 month), 6 weeks later (+/-1 month), and 12 weeks later ((+/-1 month)
  This is a 7 item questionnaire and each is scored from 0(not at all) to 4(nearly every day) for a maximum score of 21 , higher score indicating more anxiety
Change in adaptive functioning as assessed by the Adaptive Behavior Assessment System, Third Edition (ABAS-3) | baseline (+/-1 month), 6 weeks later (+/-1 month), and 12 weeks later ((+/-1 month)
  This is a 239 item questionnaire and each is scored from 0(is not able to do this behavior) to 3 [(always able to do this behavior)(or almost always)] a higher number indicating better outcome
Change in quality of life as assessed by the Autism Spectrum Quality of Life (ASQoL) questionnaire | baseline (+/-1 month), 6 weeks later (+/-1 month), and 12 weeks later ((+/-1 month)
  This is a 9 item questionnaire. Each is scored on a 4-point Likert scale from 1(not at all) to 5(totally) ,questions 6,7 and 8 are reverse scored for a maximum score range of 9-36 and higher score indicating better quality of life
Change in quality of life as assessed by the Spanish World Health Organization Quality of Life Brief Version (WHOQOL-BREF) | baseline (+/-1 month), 6 weeks later (+/-1 month), and 12 weeks later ((+/-1 month)
  This is a 26 item questionnaire ,with 4 domains. Each is scored from 1(very poor) to 5(very good) ,questions 3,4 and 26 are reverse scored for a maximum raw score of 120 and higher score indicating better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pagán, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No